CLINICAL TRIAL: NCT03055949
Title: Safety and Efficacy of an Early Rehabilitation Program in Surgical Intensive Care Unit (SICU)
Brief Title: Safety and Efficacy of an Early Rehabilitation Program in Surgical Intensive Care Unit
Acronym: ERP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Suk-Kyung, Associate professor, Asan Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AsanMC-ERP
Record Dates: First submitted 2017-01-15; First posted 2017-02-16 (Actual); Last update posted 2017-02-16 (Actual); Status verified 2017-02

CONDITIONS: ICU-acquired Weakness
Keywords: early rehabilitation; early mobilization; surgical intensive care unit

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- pre-ERP (No Intervention): A group of the surgical ICU patients who had standard care before Asan medical center developed an early rehabilitation program (ERP)
- post-ERP (Experimental): A group of the surgical ICU patients who had an early rehabilitation program (ERP) within SICU care
  Interventions: Behavioral: Early rehabilitation program

INTERVENTIONS:
Behavioral: Early rehabilitation program — The investigators evaluated patients who were admitted SICU for more than 3 days for an early rehabilitation program and delivered one of 5-stepped rehabilitation program if the patient was eligible.
  Arms: post-ERP

SUMMARY:
The purpose of this study is to determine whether an early rehabilitation program in surgical intensive care unit is safe and effective in preventing critical care illness and intensive care unit acquired weakness.

DETAILED DESCRIPTION:
Due to the complications like intensive care unit-acquired weakness, critical illness polyneuropathy and neuropsychiatric disease of critical care, many organizations focus on rehabilitation in critically ill patients' management. Despite the good outcomes from papers, there are debatable issues of method, safety and efficacy of rehabilitation. The investigators developed an early rehabilitation program (ERP) in our surgical ICU management and assessed safety and efficacy of it.

The ERP started in November 2014 in our 14-bed surgical ICU in Asan Medical Center. The investigators focused on early and 5-step rehabilitation program for patients who were admitted to SICU for at least 3 days. The investigators enrolled 69 patients (pre-ERP group) for 6 months before November 2014 and 62 patients (post-ERP group) for 6 months 1 year after the ERP started. The main measures were safety issues, delirium days, 28-d ventilator free-days, 28-d ICU free-days, hospital length of stay (LOS), ICU mortality, in-hospital mortality and 1 year mortality.

ELIGIBILITY:
Inclusion Criteria:

* patients who were admitted in SICU for at least 3 days

Exclusion Criteria:

* readmission to SICU within current hospitalization open abdomen wound patients major bone fracture patients brain death patients active bleeding patients increased intra-cranial pressure patients paraplegic patients patients or their guardians did not agree with the ERP doctor's decision (Deconditioning patients, Procedure)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2014-05; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
28-day Ventilator-free days (days) | up to 28-day
  Patients who died during the study were assigned scores of 0 for 28-day ventilator-free days.
28-day ICU-free days (days) | up to 28-day
  Patients who died during the study were assigned scores of 0 for 28-day ICU-free days

SECONDARY OUTCOMES:
Time to start rehabilitation from ICU admission (days) | up to 2 weeks
ICU delirium days (days) | up to 4 weeks
Total rehabilitation days within ICU days (days) | up to 4 weeks
ICU readmission rate (%) | up to 24 weeks
ICU mortality rate (%) | up to 24 weeks
in-hospital mortality rate (%) | up to 24 weeks
1 year mortality rate (%) | 1 year follow up from ICU admission

CONTACTS AND LOCATIONS:
Overall Officials: Suk-kyung Hong, Ph.D., Principal Investigator — Asan Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bailey P, Thomsen GE, Spuhler VJ, Blair R, Jewkes J, Bezdjian L, Veale K, Rodriquez L, Hopkins RO. Early activity is feasible and safe in respiratory failure patients. Crit Care Med. 2007 Jan;35(1):139-45. doi: 10.1097/01.CCM.0000251130.69568.87. PMID 17133183
- [Result] McWilliams D, Weblin J, Atkins G, Bion J, Williams J, Elliott C, Whitehouse T, Snelson C. Enhancing rehabilitation of mechanically ventilated patients in the intensive care unit: a quality improvement project. J Crit Care. 2015 Feb;30(1):13-8. doi: 10.1016/j.jcrc.2014.09.018. Epub 2014 Oct 2. PMID 25316527
- [Result] Morris PE, Goad A, Thompson C, Taylor K, Harry B, Passmore L, Ross A, Anderson L, Baker S, Sanchez M, Penley L, Howard A, Dixon L, Leach S, Small R, Hite RD, Haponik E. Early intensive care unit mobility therapy in the treatment of acute respiratory failure. Crit Care Med. 2008 Aug;36(8):2238-43. doi: 10.1097/CCM.0b013e318180b90e. PMID 18596631
- [Result] Schweickert WD, Pohlman MC, Pohlman AS, Nigos C, Pawlik AJ, Esbrook CL, Spears L, Miller M, Franczyk M, Deprizio D, Schmidt GA, Bowman A, Barr R, McCallister KE, Hall JB, Kress JP. Early physical and occupational therapy in mechanically ventilated, critically ill patients: a randomised controlled trial. Lancet. 2009 May 30;373(9678):1874-82. doi: 10.1016/S0140-6736(09)60658-9. Epub 2009 May 14. PMID 19446324